CLINICAL TRIAL: NCT06871709
Title: Clinical and Radiographic Evaluation of Potassium Nitrate in Polycarboxylate Versus Mineral Trioxide Aggregate in Vital Pulpotomy in Primary Molars: a Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Potassium Nitrate in Polycarboxylate Versus Mineral Trioxide Aggregate in Vital Pulpotomy in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mariam Mahmoud Salah El-Mosallamy, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vital Primary Molars Pulpotmy
Record Dates: First submitted 2025-03-04; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Vital Pulp Therapies; Pulpotomy; Pulp Disease, Dental; Pulpotomies Primary Teeth; Pulp Therapy
Keywords: Mineral Trioxide Aggregate; Potassium Nitrate; MTA; Pulpotomy; Vital Pulpotomy; Vital Pulp therapy; Primary Molars; pulp therapy; Pulp disease
MeSH Terms: conditions — Dental Pulp Diseases | interventions — potassium nitrate; Polycarboxylate Cement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Potassium Nitrate in Polycarboxylate cement) (Experimental): Potassium nitrate (KNO3) is a superior desensitizer for hypersensitive teeth. Used with polycarboxylate cement, it serves as an effective liner for deep carious lesions. Also when placed under deep restorations with less than 1 mm of protective dentin remaining, it was effective in preserving pulpal vitality and it diminished the incidence and severity of post-restoration pain. As temporary cement (Kno3/zinc oxide eugenol [ZOE]) It reduced pain following full crown preparation.
  Interventions: Combination Product: Potassium Nitrate in Polycarboxylate cement
- Group 2 (Mineral Trioxide Aggregates "MTA") (Active Comparator): Mineral trioxide aggregate (MTA) has been recommended as the gold standard for vital pulp therapy as it showed a high success rate clinically and radiographically when compared to other materials due to its biocompatibility, antibacterial properties and excellent sealing ability
  Interventions: Other: MTA-Anglus

INTERVENTIONS:
Combination Product: Potassium Nitrate in Polycarboxylate cement — The application of polycarboxylate cement containing 5% KNO3 for direct capping of traumatically exposed pulp in animal models did not result in any degenerative changes in dental pulp, thought creating optimal conditions for preservation of pulp vitality.
  Polycarboxylate cement has very thin film thickness and bonds firmly to the tooth structure, is capable of withstanding the overlying pressure during restoration procedures. The good adhesive properties of polycarboxylate cement containing 5% KNO3 guaranteed the closure of cavity, good and lasting protection of traumatically exposed dental pulp and the formation of alkaline environment possessing a strong antiacidic, anti-inflammatory and antibacterial effect of this pulp capping material, creating optimal conditions for expression of its natural reparative potential. The increased release of potassium nitrate from polycarboxylate cement by time, might be the cause of decreasing the inflammatory intensity
  Arms: Group 1 (Potassium Nitrate in Polycarboxylate cement)
Other: MTA-Anglus — Mineral Trioxide Aggregate (MTA) has been the gold standard material for primary tooth pulpotomy. MTA has antimicrobial properties, excellent sealing ability, is biocompatible and has a dentinogenic effect on pulp tissue by stimulating the release of cytokines from bone cells, which promotes hard tissue formation. Furthermore, MTA maintains pulp tissue integrity while having no cytotoxic effects. Nevertheless, the clinical application of MTA has been limited due to some properties such as its long setting time, difficulty in its handling, being washed out, discoloration, and increased cost. These urged the search for an alternative pulpotomy material to MTA
  Arms: Group 2 (Mineral Trioxide Aggregates "MTA")

SUMMARY:
The purpose of this RCT is to compare the clinical/radiographic outcomes of Potassium nitrate in polycarboxylate cement and MTA as pulpotomy biomaterials used for asymptomatic vital primary lower second molar and this will help to clinically evaluate the use of alternative material in vital pulpotomy in primary molars with deep carious cavities.

Emphasis is set on avoiding total pupectomy and maintaining radicular pulp vitality therefore maintain the tooth in a viable condition till it's shedding and eruption of the permanent successor.

DETAILED DESCRIPTION:
Introduction:

Dental caries continues to be a significant health issue, with a very high prevalence in children worldwide. For a variety of reasons (lack of proper dental education, lack of access to dental care, "silent symptomatology," etc.), treatment is frequently initiated once the progression degree has reached a deep, cavitated stage, often with pulp involvement. The primary purpose of pulp therapy in deciduous dentition is to promote the health of the teeth and their supporting tissues in order to maintain the proper functions of the oro-facial complex (mastication, speech, aesthetics), and ultimately to retain the teeth in their position to preserve arch length. Primary teeth are referred to as "the best space maintainers" as they effectively preserve space for their successors.

Carious primary teeth with normal pulp or reversible pulpitis should be treated with vital pulp procedures. Currently, three vital pulp therapy (VPT) options exist for treating deep dentin caries lesions approximating the pulp in vital primary teeth: indirect pulp treatment (IPT), direct pulp cap (DPC), and pulpotomy.

VPT is primarily recommended to be performed in young patients because of the high healing capacity of pulp tissue compared to older patients. An adequate blood supply is required to maintain the pulp's vitality. Furthermore, the presence of a healthy periodontium is required for VPT to be effective, as teeth with moderate to severe periodontal disease are not candidates for treatment. In cases with an inadequate coronal seal and subsequent bacterial microleakage, the prognosis for VPT is significantly reduced.

Pulpotomy is a conservative clinical procedure performed on pediatric patients, and most recently on adult patients too, that involves the removal of the coronal pulp while preserving the radicular pulp. The rationale is based on the healing capacity of the remaining pulp tissue following surgical amputation of the affected or infected coronal pulp. Following hemostasis, the exposed pulp is covered with either a pulp-capping agent that promotes healing or an agent to fix the underlying tissue.

Most recently, Mineral Trioxide Aggregate (MTA) has been the gold standard material for primary tooth pulpotomy. MTA has antimicrobial properties, excellent sealing ability, is bio-compatible and has a dentinogenic effect on pulp tissue by stimulating the release of cytokines from bone cells, which promotes hard tissue formation. Furthermore, MTA maintains pulp tissue integrity while having no cytotoxic effects. Nevertheless, the clinical application of MTA has been limited due to some properties such as its long setting time, difficulty in its handling, being washed out, discoloration, and increased cost. These urged the search for an alternative pulpotomy material to MTA.

Potassium Nitrate (KNO3) is an effective desensitizer for hypersensitive teeth9. Animal studies found satisfactory results using the combination of 5% KNO3 in polycarboxylate cement as a direct pulp capping material10. Clinical studies examined KNO3 in polycarboxylate as a pulp capping or pulpotomy material in vital pulp therapy.

Indirect capping with 5% KNO3 in polycarboxylate cement was compared to calcium hydroxide liner in treating reversible pulpitis in permanent teeth. The study found that 5% KNO3 in polycarboxylate cement provided effective analgesia and restored electrical excitability faster than calcium hydroxide.

A study showed that after two years of direct capping with KNO3 /dimethyl isosorbide/polycarboxylate cement in carious exposed vital pulp, all patients remained clinically and radiographically normal. Another 4-year clinical and radiographic evaluation of teeth treated with KNO3 in polycarboxylate for deep exposed and non-exposed carious lesions revealed a 97.7% success rate in the exposed group and 100% success rate in the non-exposed group.

Furthermore, on a recently published clinical study that was carried out on young immature lower first permanent molars in the Endodontic department, Faculty of dentistry, Cairo university, that was comparing KNO3 in polycarboxylate to MTA. It was revealed that KNO3 in polycarboxylate cement is a viable and cost-effective alternative to MTA for pulpotomy in immature caries-exposed permanent molars.

In conclusion, KNO3 in polycarboxylate offers low cost and easy manipulation. However, to our knowledge no randomized clinical trials (RCTs) have evaluated the use of polycarboxylate with KNO3 as a pulpotomy material for primary dentition.

Methods:

Study Setting and location

* Source of patients: this study will be conducted in the outpatient clinics of the Pediatric dentistry and Dental Public Health Department - Faculty of Dentistry, Cairo University - Egypt.
* Operator: The Principal Investigator.
* Dental units: Knight Midmark Biltmore dental unit (Midmark Corporation 1700 S. Patterson Blvd. Suite 400 Dayton, Ohio 45409, USA)
* X-ray film: Intraoral digital periapical Xray.

Intervention:

The principal investigator will carry out all treatment procedures, and the patients will be randomly assigned to any of them.

For both interventions:

1. Informed consent from participating children's parents.
2. Baseline records photographs, percussion test, periapical radiograph and personal data collection.
3. Diagnostic charts with personal, medical and dental history will be filled.
4. Allocation (concealed by withdrawing a sealed opaque envelope containing Four-folded numbered papers containing the type of dressing material that will be used then writing the patient's name and I.D. on it and will be opened after performing the access cavity).
5. Clinical examination will be performed to assess the clinical inclusion criteria. (Pulpal and periapical diagnoses are established after clinical examination).
6. Preoperative and Postoperative photographs will be taken.
7. The radiographic examination will be performed by taking a periapical x-ray using (parallel technique) to assess the inclusion criteria. The preoperative radiograph will serve as a reference for the follow-up radiographs. Standardization of the technique to avoid any distortion in the vertical dimension and to provide reproducible images using x-ray holding device.
8. Preoperative and postoperative radiographs will be taken by parallel technique using XCP film holder.
9. Administration of inferior local anesthesia at the side of the affected tooth.
10. Application of rubber dam for isolation, then a standardized pulpotomy procedure will be performed using a large sterile round end bur in a high-speed handpiece with copious irrigation, a sharp spoon excavator will remove pulpal tissues to the orifice level. Hemostasis will be achieved by the application of a wet cotton pellet. Children will then be allocated into either one of the groups alternatively depending on the pulpotomy medicament used as follows:

Group I (Experimental group) pulpotomy using KNO3 (potassium salt, Technogene Corp., Egypt) in polycarboxylate cement:

1. After complete hemostasis, 5% potassium nitrate (powder) (premixed KNO3 with zinc oxide powder (zinc oxideTm , jK Dental Vision, Egypt), 5gm to 95gm by weight) which will mixed with the polyacrylic acid (liquid) (poly zinc +, Prevest DentPro, India) in 1:1 P/L ratio will be applied using a composite applicator and gently placed over the pulp stumps then gentle condensation in the pulp chamber will be done by a moistened cotton pellet and then the rest of the pulp chamber will be filled with glass ionomer restoration (Micron Superior, Prevest DentPro, India).
2. Tooth will be restored with a stainless-steel crown (Kids Crowns, Shinhung, South Korea) cemented using glass ionomer cement (Micron Lutting, Prevest DentPro, India).

Group II (Control group) pulpotomy using MTA (Angelus, Londrina, Brazil):

1. After complete hemostasis. MTA+ saline will be manipulated in the ratio of 3:1 (powder: liquid) to obtain a putty mix. This mix will be placed over the radicular pulp with the help of a suitable sterile amalgam carrier. Gentle condensation of the mix will be done in the pulp chamber with a moistened cotton pellet, followed by the application of glass ionomer restoration (Micron Superior, Prevest DentPro, India).
2. Tooth will then be restored with a stainless-steel crown (Kids Crowns, Shinhung, South Korea) cemented using glass ionomer cement (Micron Lutting, Prevest DentPro, India).

ELIGIBILITY:
❖ Inclusion Criteria:

1. Children aged 4 to 7 years, in good general health.
2. Children with vital, deeply carious primary molars.
3. No history of spontaneous pain, pathological mobility, draining sinus tract, redness or swelling of the vestibule.
4. Normal gingival and periodontal condition, with no sensitivity to vestibular palpation, and no pain on percussion test.
5. No sign of radiolucency in periapical or furcation area.
6. No widening of PDL space or loss of lamina dura continuity.
7. No evidence of internal/external pathological root resorption.

Exclusion Criteria:

1. Children with a physical disability or medical disability.
2. Unrestorable molars.
3. Uncooperative patient.
4. Parent unable to attend Follow- up visits.
5. Parents refuse to give written informed consent.
6. If the access was opened and irreversible pulpitis was evident.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | Baseline, 1 week, 3 month, 6, 9 and 12 months after treatment
  1. Post-operative pain: will be recorded by verbal question to patient/ parent.
  2. Soft tissue pathology: will be recorded by visual clinical examination.
  3. Pain to percussion: will be recorded by percussion test (by the back of the dental mirror).
  4. Pathological mobility: will be recorded by mobility test (pressure using the end of two dental mirrors).

SECONDARY OUTCOMES:
Radiographic success rate | Baseline, 3 month, 6 and 12 months after treatment
  1. Absence of external and internal root resorption: will be recorded by using intraoral digital periapical X Ray.
  2. Absence of any pulp stones: will be recorded by using intraoral digital periapical X Ray.
  3. Absence of any furcation and periapical radiolucency: will be recorded by using intraoral digital periapical X Ray.
  4. Absence of any widening in periodontal ligament space: will be recorded by using intraoral digital periapical X Ray.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No